CLINICAL TRIAL: NCT02009059
Title: Accuracy of Non-invasive Temperature Measurement in Deep Hypothermia; a Prospective Cohort Study
Brief Title: Accuracy of Non-invasive Temperature Measurement in Deep Hypothermia
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: scs-2013
Record Dates: First submitted 2013-11-11; First posted 2013-12-11 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-01

CONDITIONS: Hypothermia
Keywords: hypothermia; Temperature; epitympanic; pre-hospital
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non-invasive temperature in hypothermia: Adult patients undergoing elective thoracic surgery in deep hypothermia
  Interventions: Device: Non-invasive temperature in hypothermia

INTERVENTIONS:
Device: Non-invasive temperature in hypothermia — accuracy of non-invasive temperature measurement in deep hypothermia compared to core temperature
  Other Names: metraux epitympanic, nasopharyngeal, 3M spotOn

SUMMARY:
In pre-hospital care, there are few non-invasive thermometers that are proved both robust and accurate. The aim of this study is to investigate the accuracy of a certain ear-canal based thermometer on patients undergoing thoracic surgery in deep hypothermia.

DETAILED DESCRIPTION:
The study is a prospective cohort study on patients undergoing elective thoracic surgery in deep hypothermia. The goal is to assess the accuracy of non-invasive temperature devices compared to a gold standard representing core temperature.

At the study hospital, Oslo University Hospital Rikshospitalet, patients undergoing thoracic surgery will already have several routes of temperature monitoring as part of standard procedure. Before cardiopulmonary bypass bladder temperature is normally used as a reference for core temperature. After cardiopulmonary bypass is established, temperature is monitored directly in the circulating blood, hence reflecting core temperature.

For measuring the epitympanic temperature we will use the Metraux Epitympanic Thermometer (Walpoth, Galdikas et al. 1994), a nasopharyngeal temperature probe (Mon-a-Therm, General Purpose Temperature Probe 12Fr/Ch, Covidien) and a new transcutaneous device (SpotOn 3M). The temperature will be measured in degrees Celsius. The first reading will be noted just after induction of anaesthesia and compared to the bladder temperature. After cardiopulmonary bypass (CPB) is established and therapeutic hypothermia is induced, the values for both non-invasive and blood temperature will be recorded every minute. After reaching the target temperature according to the blood temperature, we will continue recording the non-invasive temperature until relative similarity is established. The process will be repeated during re-warming.

ELIGIBILITY:
Inclusion Criteria:

* Adult >18 years
* Elektive cardiac surgery in deep hypothermia
* No pathology in ear canal on otoscopy

Exclusion Criteria:

* Pathology in ear canal
* non-consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective thoracic surgery in deep hypothermia
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-11 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Temperature in degrees celsius | The patients will be followed during the induced per-operative hypothermia, an expected average of 1,5 hours.
  The temperature reading from the epitympanic thermometer will be recorded every two minutes during deep hypothermia and compared to the temperature measured in the cardiopulmonary bypass circuit.

CONTACTS AND LOCATIONS:
Overall Officials: Leiv Arne Rosseland, MD, Phd, Study Director — Division of Emergencies and Critical Care, Oslo University Hospital, Oslo, Norway
Locations (1):
- Oslo University Hospital, Rikshospitalet, Oslo, Norway